CLINICAL TRIAL: NCT03569579
Title: A Randomized, Open-label, Single Dose, Crossover Study to Evaluate the Effect of D797 on Pharmacokinetics of D324 in Healthy Volunteers
Brief Title: CKD-355 Drug-drug Interaction Study (CKD-355 DDI P1)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 179DDI18002
Record Dates: First submitted 2018-06-15; First posted 2018-06-26 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Central Nervous System Diseases
MeSH Terms: conditions — Central Nervous System Diseases | interventions — Memantine; Donepezil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1(Treatment A/Treatment B) (Experimental): Period 1: Treatment A(Memantine Tab. 10mg)*2T, QD, PO.
  Period 2: Treatment B(Memantine Tab. 10mg)*2T + Donepezil Tab. 10mg)*1T, QD, PO.
  Each treatment period was separated by a washout period of at least 21 dyas.
  Interventions: Drug: Memantine Tab. 10mg; Drug: Memantine Tab. 10mg + Donepezil Tab. 10mg
- Group 1(Treatment B/Treatment A) (Experimental): Period 1: Treatment B(Memantine Tab. 10mg)*2T + Donepezil Tab. 10mg)*1T, QD, PO.
  Period 2: Treatment A(Memantine Tab. 10mg)*1T, QD, PO.
  Each treatment period was separated by a washout period of at least 21 dyas.
  Interventions: Drug: Memantine Tab. 10mg; Drug: Memantine Tab. 10mg + Donepezil Tab. 10mg

INTERVENTIONS:
Drug: Memantine Tab. 10mg — Memantine Tab. 10mg* 2T/day, QD, PO
  Other Names: Ebixa Tab. 10mg
Drug: Memantine Tab. 10mg + Donepezil Tab. 10mg — Memantine Tab. 10mg* 2T/day + Donepezil Tab. 10mg * 1T/day, QD, PO
  Other Names: Ebixa Tab. 10mg + Aricept Tab. 10mg

SUMMARY:
The purpose of this study is to evaluate a pharmacokinetic drug interaction between D797 of D324 in healthy volunteers

DETAILED DESCRIPTION:
To healthy subjects of twenty(20), following treatments are administered dosing in each period and wash-out period is a minimum of 21 days.

ELIGIBILITY:
Inclusion Criteria:

1. A healthy adult whose age is over 19 years old when visiting for initial screening test
2. Body mass index(BMI) between 17.5~30.5 kg/m^2 and the body weight must be over 55kg (Body mass index (BMI) = weight (kg) / height (m)^2)
3. A person with no congenital or chronic disease in three years, no history of symptoms in internal treatment, or no knowledge in the area
4. Due to the special characteristics of drugs, the participators must be qualified to do the clinical screening after examined through hematology test and blood chemistry analysis, urinary test, the electrocardiogram (ECG), and etc.
5. The participants must be volunteered and sign in an informed consent document proven by Chonbuk National University IRB before joining a study to show that he was given informed the purpose of tests and the special characteristics of drugs.
6. The participants must have an ability and willingness to participate throughout the entire trials

Exclusion Criteria:

1. A person who had a history or symptoms of clinically aware of blood, kidney, internal secretion, gastrointestinal, urinary system, cardiovascular, liver, mental, nercous, or allergic(except subclinical seasonal allergies that is not treated at injecion) desease.
2. Who had a gistory of gastrointestinal related disease which can be affected the drug absorption (esophageal achalasia, esophagostenosis, esophageal disease, or Crohn's disease) or surgeries (except a simple appendectomy or herniotomy)
3. Who had following results after examination

   a. ALT or AST > twice higher than normal value
4. Who constantly intake 210 g/week of alcohol within 6 months of the screening. (a cup of beer (5%) (250 mL) = 10 g, a shot of soju (20%) (50mL) = 8 g, a glass of wine (!2%) (125 mL) = 12g)
5. Who participated other clinical test or took testing bioequivalence drugs in 3 months before the first clinical drug trial.
6. Whose blood pressure < 100 or ≥140(systolic blood pressure) or < 70 or ≥ 90(diastolic blood pressure)
7. Who had a medical history of alcohol and drug abuses.
8. Who had taken a drug that has a control of metabolic rate (activatioh or inhibithion) in 30 days before the first taking of clinical testing durg.
9. Who smokes more than 10 eigarettes per day.
10. Who took prescribed drugs or over-the-conuter durgs in 10 days before taking of very first clinical testing drug.
11. Who participated in whole blood donation in 2 months before the first taking of clinical testing drugs or platelet donations in 1 month before the first taking to clinical testing drugs.
12. Who has a potent to increase a danger by participating in the clinical trials or sho can interrupt interpretin test results by having serious or chronic medical and mental status or having issues in results of the screening examination.
13. Who has a histroy of an extreme sensitivity of drugs that contain donepezil hydrochloride, piperidine derivatives, memantine hydrochloride drugs.

    Who has a serious heart failure or a congestive heart failure that must be drug-treated
14. Who has a Pregnant or potentially pregnant.
15. Who has Galactose intolerance, LAPP lactose intolerance, glucose-galactose malabsorption or genetic disorders.
16. A patient with severe hepatopathy
17. A patient with moderate nephropathy.
18. A person who is not determined unsuitable to participate in this test by the researchers.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2018-05-21 (Actual); Study Completion 2018-06-04 (Actual)

PRIMARY OUTCOMES:
AUCt of Memantine | 1Day 0h, 1h, 2h, 3h, 4h, 5h, 6h, 7h, 8h, 12h, 24h, 48h, 72h, 120h, 168h, 216h
  Area under the plasma concentration of Memantine versus time curve from time zero to time of last quantifiable concentration
Cmax of Memantine | 1Day 0h, 1h, 2h, 3h, 4h, 5h, 6h, 7h, 8h, 12h, 24h, 48h, 72h, 120h, 168h, 216h
  Maximum plasma concentration of Memantine

SECONDARY OUTCOMES:
AUCinf of Memantine | 1Day 0h, 1h, 2h, 3h, 4h, 5h, 6h, 7h, 8h, 12h, 24h, 48h, 72h, 120h, 168h, 216h
  Area under the plasma concentration of Memantine versus time curve from time zero to time infinity
Tmax of Memantine | 1Day 0h, 1h, 2h, 3h, 4h, 5h, 6h, 7h, 8h, 12h, 24h, 48h, 72h, 120h, 168h, 216h
  Time to maximum concentration of of Memantine
t1/2 of Memantine | 1Day 0h, 1h, 2h, 3h, 4h, 5h, 6h, 7h, 8h, 12h, 24h, 48h, 72h, 120h, 168h, 216h
  Apparent terminal half-life of Memantine
CL/F of Memantine | 1Day 0h, 1h, 2h, 3h, 4h, 5h, 6h, 7h, 8h, 12h, 24h, 48h, 72h, 120h, 168h, 216h
  Total body clearance of Memantine
Vd/F of Memantine | 1Day 0h, 1h, 2h, 3h, 4h, 5h, 6h, 7h, 8h, 12h, 24h, 48h, 72h, 120h, 168h, 216h
  Apparent volume of distribution of Memantine

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Ho Jang, Professor, Principal Investigator — Chonbuk National University Hospital
Locations (1):
- Chonbuk National University Hospital, Jeonju, South Korea